CLINICAL TRIAL: NCT03160742
Title: Pilot Study of a Non-Invasive Central Venous Pressure Monitoring System in Children
Status: Terminated | Type: Observational
Why Stopped: Study device is incorrect size for pediatric patients
Sponsor: Boston Children's Hospital (Other)
Collaborators: Mespere Lifesciences Inc. (Industry)
Responsible Party: Principal Investigator, Kirsten Odegard, Cardiac Anesthesiologist, Boston Children's Hospital
Other Study IDs: IRB-P00024295
Record Dates: First submitted 2017-05-18; First posted 2017-05-19 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Central Venous Pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Non-invasive monitoring: In addition to standard monitoring, the Mespere VENUS 200CVP system will be used to record central venous pressures.
  Interventions: Device: Mespere VENUS 200CVP system

INTERVENTIONS:
Device: Mespere VENUS 200CVP system — Non-invasive sensor placed on the neck

SUMMARY:
The goal of this research study is to determine the feasibility and accuracy of Mespere Life Science non-invasive central venous pressure monitoring system (Mespere VENUS 2000CVP system) in children with congenital heart disease (CHD).

DETAILED DESCRIPTION:
Central venous pressure (CVP), also known as right atrial pressure (RAp), is a reflection of the right heart filling pressure i.e the preload of the right ventricle. Assessment of the CVP is essential in the management of different clinical situations in children. Invasive CVP monitoring by placement of a CVP catheter either in the internal jugular vein or the subclavian vein is the gold standard way of measuring the CVP both in children and adults. However, placing a CVP catheter in a child can be challenging, time consuming, often requires the child to be sedated and it is not without complications.

Being able to reliably measure the CVP noninvasively would be of great benefit for sick children as it may allow diagnoses to be made quickly and help guide treatment.

The goal of this proposal is to determine the feasibility and accuracy of Mespere Life Science non-invasive central venous pressure monitoring system (Mespere VENUS 2000CVP system) in children with congenital heart disease (CHD).

ELIGIBILITY:
Inclusion Criteria:

* 12 months of age to 10.9 years of age
* Scheduled to undergo a cardiac surgery with central venous pressure catheter monitoring at Boston Children's Hospital

Exclusion Criteria:

* undergo a procedure that does not require a central venous pressure catheter as part of routine monitoring
* Have a known venous occlusion or any other reason the central venous pressure may be unreliable
* Allergy to medical grade adhesives or have any pre-existing skin irritation/eczema at the sensor site
* Emergently scheduled procedures

Ages: 12 Months to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 30 children ages 12 months to 10.9 years scheduled to undergo a cardiac surgery with central venous pressure catheter monitoring at Boston Children's Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2018-04-25 (Actual); Primary Completion 2018-04-25 (Actual); Study Completion 2018-09-14 (Actual)

PRIMARY OUTCOMES:
Accuracy of Mespere VENUS 2000CVP | The data will be collected for the length of the cardiac surgery, up to 6 hours.
  The correlation between the non-invasive measurements from the Mespere VENUS 2000CVP system and the invasive central venous pressure measurements that are continuously collected as standard of care.

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Odegard, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No